CLINICAL TRIAL: NCT01919255
Title: Evaluation of PICOLIGHT Plus COOLPREP, PICOLIGHT Plus CLICOLON for Bowel Preparation (The Phase II Prospective Randomized Clinical Trial)
Brief Title: Evaluation of PICOLIGHT Plus COOLPREP, PICOLIGHT Plus CLICOLON for Bowel Preparation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Dae Kyung Sohn, MD., PHD, Center for Colorectal Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NCC-CAN-001
Record Dates: First submitted 2013-08-03; First posted 2013-08-08 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Colonoscopy; Bowel preparation; Picolight; Clicolon; Coolprep
MeSH Terms: interventions — Magnesium Oxide; picosulfate sodium; sodium sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Picolight + Coolprep (Day-Prior) (Active Comparator): Picolight (1p/250cc, 5PM) + Coolprep (500cc x 2, 8PM)[Day-Prior]
  Interventions: Drug: Picolight + Coolprep
- Picolight + Clicolon (Day-Prior) (Active Comparator): Picolight (1p/250cc, 5PM) + Clicolon (4T x 4, 8PM) [Day-Prior]
  Interventions: Drug: Picolight + Clicolon
- Picolight + Coolprep (Split-Dose) (Active Comparator): Picolight (1p/250cc, 7PM) + Coolprep (500cc x 2, 5AM)[Split-Dose]
  Interventions: Drug: Picolight + Coolprep
- Picolight + Clicolon (Split-Dose) (Active Comparator): Picolight (1p/250cc, 7PM) + Clicolon (4T x 4, 5AM)[Split-Dose]
  Interventions: Drug: Picolight + Clicolon

INTERVENTIONS:
Drug: Picolight + Coolprep — Picolight (1p/250cc, 5PM) + Coolprep (500cc x 2, 8PM)[Day-Prior] Picolight (1p/250cc, 7PM) + Coolprep (500cc x 2, 5AM)[Split-Dose]
  Other Names: Picolight(Citric acid, Magnesium Oxide, Sodium picosulfate); Coolprep(PEG 3350 + EL, Ascobic acid, Sodium sulfate)
  Arms: Picolight + Coolprep (Day-Prior); Picolight + Coolprep (Split-Dose)
Drug: Picolight + Clicolon — Picolight (1p/250cc, 5PM) + Clicolon (4T x 4, 8PM) [Day-Prior] Picolight (1p/250cc, 7PM) + Clicolon (4T x 4, 5AM)[Split-Dose]
  Other Names: Picolight(Citric acid, Magnesium Oxide, Sodium picosulfate); Clicolon(Sodium phosphate)
  Arms: Picolight + Clicolon (Day-Prior); Picolight + Clicolon (Split-Dose)

SUMMARY:
The purpose of this study to bowel cleansing evaluation of mixed two other type bowel preparation drug(PICOLIGHT plus COOLPREP, PICOLIGHT plus CLICOLON).

DETAILED DESCRIPTION:
To evaluate mixed-drug bowel preparation methods for decreasing side effect and increasing compliance

Picolight + Coolprep [Day-Prior] Picolight + Clicolon [Day-Prior] Picolight + Coolprep [Split-Dose] Picolight + Clicolon [Split-Dose]

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years of age
* Elective colonoscopy of outpatients(consent to the study)

Exclusion Criteria:

* Active enteritis, enteric bleeding, obstruction
* Pregnant or lactating women
* Severe liver or renal insufficiency
* Allergic to any preparation components
* History of heart disease (ischemic heart disease, congestive heart failure, arrythmia)
* History of colorectal surgery
* History abdominal surgery within 6 month
* Toxic colitis or megacolon
* Nausea or vomiting
* Status emergent abdominal surgery (ex. acute appendicitis)
* Uncontrolled clinically significant pre-existing electrolyte disturbance
* Dehydration
* Phenylketonuria
* Glucose-6-phosphate dehydrogenase deficiency
* Ileus
* Suspicious hyperphosphatemia
* Acute phosphate nephropathy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Bowel preparation quality | the day of colonoscopy
  Aronchick bowel preparation score;
  Excellent: small volume of clear liquid or greater than 95% of surface seen
  Good: large volume of clear liquid 5% to 25% of the surface but greater than 90% of surface seen
  Fair: some semi-solid stool that could be suctioned or washed away, but greater than 90% of surface seen
  Poor: semi-solid stool that could not be suctioned or washed away and less than 90% of surface seen
  Inadequate: re-preparation needed
  (* 'success' of bowel preparation is defined as Aronchick's 'Excellent' or 'Good'.)

SECONDARY OUTCOMES:
Patient tolerance | the day of colonoscopy
  Patient's tolerance;
  1= "none"; 2= "mild"; 3= "bothersome"; 4= "distressing"; 5= "severely distressing"

OTHER OUTCOMES:
Adenoma detection rate | The day of colonoscopy
  Adenoma detection rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Dae Kyung Sohn, Principal Investigator — NCC,Korea
Locations (1):
- Dae Kyung Sohn, Goyang-si, Gyeonggi-do, South Korea